CLINICAL TRIAL: NCT04129762
Title: Effect of a Diet Without Non-caloric Sweeteners on Gastrointestinal Symptoms in Patients With Irritable Bowel Syndrome and Dyspepsia
Brief Title: Effect of a Diet Without Non-caloric Sweeteners on Gastrointestinal Symptoms in Patients With IBS and Dyspepsia
Acronym: IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Nallely Bueno Hernández, Investigator In Medical Science B, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DI/19/301/03/020
Record Dates: First submitted 2019-10-08; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: IBS - Irritable Bowel Syndrome; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases | interventions — Diet; Zinostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Diet without NCS in irritable bowl syndrome (Experimental): Participants with irritable bowl syndrome are assigned to a 5 meals divided diet. In which it does not contain any products with NCS
  Interventions: Other: Diet without NCS
- Diet with NCS in irritable bowl syndrome (Active Comparator): Participants with irritable bowl syndrome are assigned to a 5 meals divided diet. In which it contain any products with NCS
  Interventions: Other: Diet with NCS
- Diet without NCS in dyspepsia (Experimental): Participants with dyspepsia are assigned to a 5 meals divided diet. In which it does not contain any products with NCS
  Interventions: Other: Diet without NCS
- Diet with NCS in dyspepsia (Active Comparator): Participants with dyspepsia are assigned to a 5 meals divided diet. In which it contain any products with NCS
  Interventions: Other: Diet with NCS

INTERVENTIONS:
Other: Diet without NCS — A standard diet in terms of macronutrients will be calculated.
  * 55% Carbohydrates
  * 20% protein
  * 25% Lipids The energy calculation will be done with the Harris Benedict formula and a diet with equivalents will be made and then a menu distributed in 5 meals, lasting 7 days.
  The menu will not contain products with NCS.
  Other Names: Diet
  Arms: Diet without NCS in dyspepsia; Diet without NCS in irritable bowl syndrome
Other: Diet with NCS — A standard diet in terms of macronutrients will be calculated.
  * 55% Carbohydrates
  * 20% protein
  * 25% Lipids The energy calculation will be done with the Harris Benedict formula and a diet with equivalents will be made and then a menu distributed in 5 meals, lasting 7 days.
  The menu will contain products with NCS.
  Other Names: Diet
  Arms: Diet with NCS in dyspepsia; Diet with NCS in irritable bowl syndrome

SUMMARY:
Digestive Functional Disorders (DFD), represent 50% of medical check ups, the symptoms interfere with patients quality of life and generate high health costs. On the other hand, with the worldwide overweight and obesity increase,causing an over production of low-calorie products, which increase the non-caloric sweeteners (NCS) consumption.

Hypothesis: A diet without NCS will reduce gastrointestinal symptoms in volunteers with dyspepsia and IBS.

Objective: To asses the effect of a diet without NCS, on the gastrointestinal symptoms in patients with dyspepsia and IBS.

Secondary Objectives: To compare the effect of a diet without NCS against a diet with NCS on anthropometry, changes in body composition, biochemical parameters, glucose and insulin. To asses the change in the gut microbiota using real-time PCR (polymerase chain reaction)

Methodology: it will be an experimental, open, parallel, controlled study lasting 12 weeks, patients with dyspepsia or IBS will be randomized assigned to a diet with or without NCS.

Laboratory studies, dietary and symptoms questionnaires, anthropometry measurements and faecal sample will be carried out.

Analysis Results: A double data capture will be carried out to minimize errors, for the statistical analysis of using the Statistical Package for the Social Sciences (SPSS) version 25, descriptive statistics will be used to report the baseline data of the volunteers. Using means and standard deviation, the variables of gastrointestinal symptoms will be used a chi-square test and a p <0.05 will be considered significant. Different analyzes will be done to evaluate volunteers with IBS and those with dyspepsia. For the intestinal microbiota analysis, a comparison will be made between the percentages of Firmicutes, Bacteroidetes and Actinobacteria of sample 1 and 2 and a chi-square test will be performed considering a p <0.05 significant

DETAILED DESCRIPTION:
Recruitment will be carried out in the gastroenterology service, where patients will have their diagnosis of IBS or dyspepsia, participants are invited to participate in the study to subsequently sign the informed consent.

Once signed the patient is scheduled for blood studies, their nutritional evaluation will be carried out and their menu will be delivered.

Patients will be followed for 12 weeks to re-conduct their nutritional evaluation and laboratory studies.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes from 18 to 65 years old
* Diagnosis of IBS or Dyspepsia
* Patients with dyspepsia must have endoscopy
* Normal or overweight BMI (18.5 - 29.9 kg / m2)
* Not suffering from chronic non-communicable or infectious diseases
* Follow the meal plan that is being given.
* Do not consume alcoholic beverages
* No Smoking
* Signing of the informed consent letter expressing your desire to participate as volunteers in the study

Exclusion Criteria:

* People who at the time of their selection are studying with acute illness of any kind
* Type 1 or 2 diabetes.
* Diagnosis of malabsorption syndrome
* Neoplasia
* Inflammatory bowel disease
* Medicine that affects the gastrointestinal tract
* Women who at the time of their selection are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The diet without NCS will change the frequency of gastrointestinal symptoms in patients with IBS. | 12 weeks
  Using ROME III criteria, the frequency of patients who present with gastrointestinal symptoms is monitored.
The diet without NCS will change the frequency of gastrointestinal symptoms in patients with dyspepsia. | 12 weeks
  Using ROME III criteria, the frequency of patients who present with gastrointestinal symptoms is monitored.

SECONDARY OUTCOMES:
The changes in the weight of the patients with irritable bowel syndrome, from the beginning of the diet, at 6 weeks and at 12 weeks | at the week 1, 6 and 12
  For the evaluation we are going to use weight in kilograms
The changes in the weight of the patients with dyspepsia, from the beginning of the diet, at 6 weeks and at 12 weeks | at the week 1, 6 and 12
  For the evaluation we are going to use weight in kilograms
The changes in the body composition in patients with irritable bowel syndrome, from the beginning of the diet, at 6 weeks and at 12 weeks | at the week 1, 6 and 12
  We are going to use RJL system IV for body composition we will report the changes in percentage of water, fat and muscle.
The changes in the body composition in patients with dyspepsia, from the beginning of the diet, at 6 weeks and at 12 weeks | at the week 1, 6 and 12
  We are going to use RJL system IV for body composition we will report the changes in percentage of water, fat and muscle.
The changes in the waist circumference in patients with irritable bowel syndrome, from the beginning of the diet, at 6 weeks and at 12 weeks | at the week 1, 6 and 12
  For the evaluation we are going to use waist circumference in centimeters
The changes in the waist circumference in patients with dyspepsia, from the beginning of the diet, at 6 weeks and at 12 weeks | at the week 1, 6 and 12
  For the evaluation we are going to use waist circumference in centimeters
The changes in glucose in the patients with irritable bowel syndrome, from the beginning and end of the diet | at the week 1 and 12
  For the changes we are going to use glucose in mg / dl
The changes in glucose in the patients with dyspepsia, from the beginning and end of the diet | at the week 1 and 12
  For the changes we are going to use glucose in mg / dl
The changes insulin in the patients with irritable bowel syndrome, at the beginning and end of the diet | at the week 1 and 12
  For the serological changes in the insulin we are going to use the measure in IU
The changes insulin in the patients with dyspepsia, at the beginning and end of the diet | at the week 1 and 12
  For the serological changes in the insulin we are going to use the measure in IU
The changes in the lipids profile in the patients with irritable bowel syndrome, at the beginning and end of the diet | at the week 1 and 12
  For the serological changes in the lipid profile we are going to use triglycerides in mg/dl, total cholesterol in mg/dl, HDL in mg/dl, cholesterol, LDL in mg / dl.
The changes in the lipids profile in the patients with dyspepsia, at the beginning and end of the diet. | at the week 1 and 12
  For the serological changes in the lipid profile we are going to use triglycerides in mg/dl, total cholesterol in mg/dl, HDL in mg/dl, cholesterol, LDL in mg / dl.
Effect of the diet without NCS in gut microbiota in patients with irritable bowel syndrome at the beginning and end of the diet | at the week 1 and 12
  Using real-time PCR, the effect of the diet without NCS, on the gut microbiota of patients with irritable bowel syndrome
Effect of the diet without NCS in gut microbiota in patients with dyspepsia at the beginning and end of the diet | at the week 1 and 12
  Using real-time PCR, the effect of the diet without NCS, on the gut microbiota of patients with dyspepsia

CONTACTS AND LOCATIONS:
Locations (1):
- Nallely Hernandez Bueno, Mexico City, Cuauhtemoc, Mexico